CLINICAL TRIAL: NCT00833170
Title: Pediatric Inflammatory Bowel Disease Collaborative Research Group Registry
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey Hyams, MD, Study Principal Investigator, Connecticut Children's Medical Center
Other Study IDs: PIBDCRG1
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Disease
Keywords: pediatric inflammatory bowel disease; multiple site study
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Pediatric Inflammatory Bowel Disease Collaborative Research Group Registry is to study the contemporary natural history of children <16 years of age newly diagnosed with inflammatory bowel disease. The project follows these children quarterly from diagnosis examining clinical, laboratory, and humanistic outcomes. Genetic and serologic monitoring is performed on the study population.

DETAILED DESCRIPTION:
Observations of children with IBD often suggest a more severe course than that found in adults. Explanations for this are unclear, especially since children are less likely to engage in some behaviors (e.g., smoking) that may have a deleterious effect on disease course as noted in adults. In many ways children are a better "experimental model" of IBD because they don't have as many confounding medical factors as adults. Both Crohn's disease and ulcerative colitis are believed to result from a complex interaction of genetic and environmental factors (1). Recently, the gene CARD15/NOD2 on chromosome 16 has been identified in approximately 25% of Caucasian patients with Crohn's disease and is felt to be a significant predisposing factor to the development of fibrostenosing disease (2). Additionally, seropositivity for perinuclear antinuclear cytoplasmic factor (pANCA) has been demonstrated much more frequently in patients with ulcerative colitis than in those with Crohn's disease, while anti-Saccharomyces antibody (ASCA) is more common in the latter population (3). The importance of these serological abnormalities is not clear, though some data suggest an influence on the development of complications.

Our hypothesis is that phenotypic, genotypic and serologic characteristics may provide prognostic information on response to therapy and course in children with IBD. This type of prognostic information is particularly important as newer therapies are developed.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of ulcerative colitis, Crohn's disease, indeterminate colitis
2. Age up to 16 years and zero days at time of diagnosis
3. Informed consent/assent from parent/guardian and patient
4. Ability to be available for regular follow-up visits

Exclusion Criteria:

1. Diagnosis of IBD greater than 1 month prior to presentation to participating center
2. Age greater than 16 years and zero days
3. Inability to be available for regular follow-up visits

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children <16 years old with inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2002-01-28 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Clinical activity following biologic and immunomodulatory therapy | 10 years
  Clinical Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Hyams, M.D., Principal Investigator — Connecticut Children's Medical Center
Locations (28):
- United States (24):
  - University of Alabama, Birmingham, Alabama
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Childrens Hospital, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - The John's Hopkins Medical Institute, Baltimore, Maryland
  - Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Steven & Alexandra Cohen Children's Medical Center, New Hyde Park, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Children's Hospital At Montefiore, The Bronx, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Medical Center, Dayton, Ohio
  - Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - IWK Health Centre,, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine Hospital, Montreal, Quebec